CLINICAL TRIAL: NCT01570192
Title: Impact of Aggressive Empiric Antibiotic Therapy and Duration of Therapy on the Emergence of Antimicrobial Resistance During the Treatment of Hospitalized Subjects With Pneumonia Requiring Mechanical Ventilation
Brief Title: Clinical Trials to Reduce the Risk of Antimicrobial Resistance
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: NIAID terminated the study due to low subject enrollment
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-0060
Record Dates: First submitted 2012-03-22; First posted 2012-04-04 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Bacterial Pneumonia
Keywords: gram negative pathogens; Pseudomonas aeruginosa; Acinetobacter; HCAP; VABP; HABP
MeSH Terms: conditions — Pneumonia, Bacterial; Pseudomonas Infections | interventions — Meropenem; Tobramycin; Linezolid; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is an open-label study with 1:1 randomization between two active treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV meropenem; parenteral aminoglycoside (Experimental): Subjects assigned to this group will receive:
  * IV meropenem (2 g infused over 3 hrs q 8 hr);
  * a parenteral aminoglycoside (tobramycin or gentamicin-5mg/kg IV Q24h or amikacin 20 mg/kg IV Q24h)
  * tobramycin nebulization
  Linezolid or vancomycin (per institutional guidelines) will be available for MRSA coverage to treat potential Gram-positive pathogens.
  Interventions: Drug: IV meropenem; Drug: Parenteral aminoglycoside; tobramycin for injection USP OR gentamicin sulfate injection solution concentrate 5mg.kg IV q24h; amikacin sulfate injection USP 20 mg/kg IV q24h; Drug: Linezolid or Vancomycin (per institutional guidelines) will be available for MRSA coverage.; Device: tobramycin nebulization
- I.V. Meropenem (Active Comparator): Subjects assigned to this group will receive IV meropenem (2 g infused over 3 hrs q 8 hr).
  Linezolid or vancomycin (per institutional guidelines) will be available for MRSA coverage to treat Gram-positive pathogens.
  **NOTE: Empiric MRSA coverage is allowed in both arms. This therapy is advised for any subjects with known or suspected MRSA entering the study. Once microbiologic results are available, this coverage may be discontinued at the investigator's discretion.
  Interventions: Drug: I.V. Meropenem; Drug: Linezolid or Vancomycin (per institutional guidelines) will be available for MRSA coverage.

INTERVENTIONS:
Drug: IV meropenem — Subjects assigned to this group will receive IV meropenem (2 g infused over 3 hrs q 8 hr).
  Other Names: Merrem I.V.
  Arms: IV meropenem; parenteral aminoglycoside
Drug: I.V. Meropenem — Subjects assigned to this group will receive IV meropenem (2 g infused over 3 hrs q 8 hr).
  Linezolid or vancomycin (per institutional guidelines) will be available for MRSA coverage
  Other Names: Merrem I.V.
  Arms: I.V. Meropenem
Drug: Parenteral aminoglycoside; tobramycin for injection USP OR gentamicin sulfate injection solution concentrate 5mg.kg IV q24h; amikacin sulfate injection USP 20 mg/kg IV q24h — a parenteral aminoglycoside (tobramycin or gentamicin-5mg/kg IV Q24h or amikacin 20 mg/kg IV Q24h)
  Arms: IV meropenem; parenteral aminoglycoside
Drug: Linezolid or Vancomycin (per institutional guidelines) will be available for MRSA coverage. — Linezolid or vancomycin (per institutional guidelines) will be available for MRSA coverage.
Device: tobramycin nebulization — tobramycin nebulization 600mg/day
  Arms: IV meropenem; parenteral aminoglycoside

SUMMARY:
The primary objective of this study is to demonstrate a low rate of emergence of antibiotic resistance in P. aeruginosa and Acinetobacter spp during the treatment of hospitalized patients with pneumonia requiring mechanical ventilation treated with PD optimized meropenem administered as a prolonged infusion in combination with a parenteral aminoglycoside plus tobramycin by inhalation (Group 1) compared to therapy with meropenem alone (Group 2 - control arm).

DETAILED DESCRIPTION:
The goal of this clinical study is to demonstrate that the application of pharmacodynamic dosing principles to the antibiotic treatment of hospitalized subjects with culture-documented pneumonia (including HABP, VABP and HCAP) requiring mechanical ventilation can inhibit the emergence of antibiotic-resistant organisms during treatment and therefore may improve the rate of a satisfactory clinical response. Antibiotic resistance is defined as an increase in meropenem or aminoglycoside MIC by two tube dilutions (fourfold) from baseline. In animal models of infection, the pharmacodynamic driver for bactericidal effect by β lactam antibiotics such as meropenem is the proportion of the dosing interval during which plasma drug levels are maintained above the MIC of the causative pathogen. The hypothesis of this study is that prolongation of time above MIC by increasing total meropenem dose and the duration of infusion will counter-select for the emergence of antimicrobial resistance during the treatment of hospitalized subjects with pneumonia (i.e. HABP, VABP and HCAP) caused by P.aeruginosa, Acinetobacter species (spp), or other pathogens with intermediate susceptibility to meropenem, and that the addition of parenteral aminoglycosides (amikacin, tobramycin or gentamicin) and nebulized aminoglycoside (tobramycin) given along optimal pharmacodynamic principles will further reduce the likelihood of resistance emergence, particularly among the non-fermenting Gram-negative bacilli, such as Pseudomonas aeruginosa and Acinetobacter spp. The observed incidence of resistance emergence to meropenem will be compared across therapeutic regimens.

ELIGIBILITY:
Inclusion criteria:

Written informed consent by the subject/subject's LAR.

Hospitalized males or females ≥ 18 yrs with respiratory failure requiring mechanical ventilation and clinical suspicion of HABP, HCAP or VABP.

Onset or exacerbation of pneumonia at least 48 hours after admission to any patient health care facility or onset of pneumonia in a nursing home or rehabilitation facility with subsequent transfer to an acute care facility

Women of childbearing potential if their pregnancy test is negative

Subjects who have received previous antibacterial therapy within 14 days of pre-treatment bronchoscopy entry may be entered only if the subject has not responded clinically.). While less than 24 hours of pre-treatment antibiotics is preferential, recovery of >104 CFU/ml in the quantitative Bronchoscopic BAL will be seen as primary evidence that the prior therapy was not efficacious and enrollment will be allowed.)

Patients should have clinical findings that support a diagnosis of HABP/VABP/HCAP:

Within 48 hours before starting empiric therapy a subject's chest radiograph should show the presence of a NEW or progressive infiltrate, cavitation, or effusion suggestive of pneumonia

Within 36 hours before the start of empiric study therapy, a quantitative culture of Bronchoscopic BAL fluid must be obtained.

Patients with VABP should have a Clinical Pulmonary Infection Score of >/= 5.

Exclusion Criteria:

Subjects with pneumonia caused by pathogens resistant to meropenem (MIC greater than or equal to 16µg/ml) or a prior meropenem therapy failure.

Subjects with contra-indications to ANY study medication, in particular with known or suspected allergy or hypersensitivity.

Women who are pregnant or lactating.

Subjects taking anticonvulsant medications for a known seizure disorder.Patients with a history of seizures, AND who are stabilized on anti-seizure medication, may be enrolled into the study at the discretion of the site investigator.

Subjects with known or suspected community acquired bacterial pneumonia (CABP) or viral pneumonia; or Subjects with acute exacerbation of chronic bronchitis without evidence of pneumonia.

Subjects with primary lung cancer or another malignancy metastatic to the lungs.

Subjects who were previously enrolled in this study.

Subjects who have had an investigational drug or have used an investigational device within 30 days prior to entering the study.

Subjects with another focus of infection requiring concurrent antibiotics that would interfere with evaluation of the response to study drug.

Subjects with cystic fibrosis, AIDS with a CD4 lymphocyte count <200 cells/µl, neutropenia (absolute neutrophil count <500 cells/ml), known or suspected active tuberculosis.

Subjects with little chance of survival for the duration of study therapy.

Subjects with an APACHE II score >35.

Subjects with underlying condition(s) which would make it difficult to interpret response to the study drugs.

Subjects with hypotension or acidosis despite attempts at fluid resuscitation. Subjects requiring ongoing treatment with vasopressors will be eligible for the study if their hypotension is controlled and acidosis has resolved. Subjects with intractable septic shock are not eligible for enrollment.

Subjects who have undergone bone marrow transplantation.

Subjects with profound hypoxia as defined by a PaO2/FiO2 ratio <100.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George L Drusano, MD, Principal Investigator — University of Florida
Locations (11):
- United States (8):
  - InClin, Inc., San Mateo, California
  - UFL Department of Medicine: Pulmonary, Critical Care and Sleep Medicine, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - JMI Laboratories, North Liberty, Iowa
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Weill Cornell Medical Center of Cornell University, New York, New York
  - Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
- Institut de Cardiologie, Groupe Hospitalier Pitie-Salpetriere, Paris, France
- Hannover Clinical Trial Center GmbH, Hanover, Germany
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hospital-acquired pneumonia in adults: diagnosis, assessment of severity, initial antimicrobial therapy, and preventive strategies. A consensus statement, American Thoracic Society, November 1995. Am J Respir Crit Care Med. 1996 May;153(5):1711-25. doi: 10.1164/ajrccm.153.5.8630626. No abstract available.
- [Background] Bauernfeind A, Jungwirth R. In Vitro Activity of SM 7338 and Imipenem. 28th ICAAC, Los Angeles, October 1988. Abstract 599
- [Background] Calandra GB, Hesney M, Brown KR. Imipenem/cilastatin therapy of serious infections: a U.S. multicenter noncomparative trial. Clin Ther. 1985;7(2):225-38. PMID 3886144
- [Background] Clarke AM, Zemcov SJV. SM 7338 (ICI 194,660), A New DHP-1 Stable Carbapenem; In Vitro Activity Against a Wide Range of Canadian Clinical Isolates. 28th ICAAC, Los Angeles, October 1988. Abstract 598.
- [Background] Craig WA. Pharmacokinetic/pharmacodynamic parameters: rationale for antibacterial dosing of mice and men. Clin Infect Dis. 1998 Jan;26(1):1-10; quiz 11-2. doi: 10.1086/516284. PMID 9455502
- [Background] Craig WA. The pharmacology of meropenem, a new carbapenem antibiotic. Clin Infect Dis. 1997 Feb;24 Suppl 2:S266-75. doi: 10.1093/clinids/24.supplement_2.s266. PMID 9126702
- [Background] Dandekar PK, Maglio D, Sutherland CA, Nightingale CH, Nicolau DP. Pharmacokinetics of meropenem 0.5 and 2 g every 8 hours as a 3-hour infusion. Pharmacotherapy. 2003 Aug;23(8):988-91. doi: 10.1592/phco.23.8.988.32878. PMID 12921245
- [Background] Data on file. Drug Development Department, AstraZeneca Pharmaceuticals, Wilmington,DE 19897.
- [Background] Drusano GL. Prevention of resistance: a goal for dose selection for antimicrobial agents. Clin Infect Dis. 2003 Jan 15;36(Suppl 1):S42-50. doi: 10.1086/344653. PMID 12516029
- [Background] Drusano GL, Liu W, Fregeau C, Kulawy R, Louie A. Differing effects of combination chemotherapy with meropenem and tobramycin on cell kill and suppression of resistance of wild-type Pseudomonas aeruginosa PAO1 and its isogenic MexAB efflux pump-overexpressed mutant. Antimicrob Agents Chemother. 2009 Jun;53(6):2266-73. doi: 10.1128/AAC.01680-08. Epub 2009 Mar 16. PMID 19289521
- [Background] Edwards JR, Wannop C. SM 7338, A New Carbapenem Antibacterial: In Vitro Activity Against Imipenem-Resistant Ps. aeruginosa. 27th ICAAC, New York October 1987, Abstract 754.
- [Background] Edwards JR, Turner PJ, Withnell ES, et al. SM 7338, A New Carbapenem Antibacterial: In Vitro Activity Against Bacterial Strains of Clinical Origins. 27th ICAAC, New York, October 1987, Abstract 755.
- [Background] Edwards JR, Turner PJ, Wannop C, Withnell ES, Grindey AJ, Nairn K. In vitro antibacterial activity of SM-7338, a carbapenem antibiotic with stability to dehydropeptidase I. Antimicrob Agents Chemother. 1989 Feb;33(2):215-22. doi: 10.1128/AAC.33.2.215. PMID 2655530
- [Background] Fagon JY, Chastre J, Novara A, Medioni P, Gibert C. Characterization of intensive care unit patients using a model based on the presence or absence of organ dysfunctions and/or infection: the ODIN model. Intensive Care Med. 1993;19(3):137-44. doi: 10.1007/BF01720528. PMID 8315120
- [Background] Fink MP, Snydman DR, Niederman MS, Leeper KV Jr, Johnson RH, Heard SO, Wunderink RG, Caldwell JW, Schentag JJ, Siami GA, et al. Treatment of severe pneumonia in hospitalized patients: results of a multicenter, randomized, double-blind trial comparing intravenous ciprofloxacin with imipenem-cilastatin. The Severe Pneumonia Study Group. Antimicrob Agents Chemother. 1994 Mar;38(3):547-57. doi: 10.1128/AAC.38.3.547. PMID 8203853
- [Background] Fukasawa M, Sumita Y, Tada E, et al. SM 7338, A New Carbapenem Antibacterial: In Vitro Activity Against 1607 Clinical Strains of Gram-Positive and Gram-Negative Pathogens. 27th ICAAC, New York, October 1987, Abstract 753.
- [Background] Fukasawa M, Tada E, Nouda H, et al. Induction and Inhibition of b-Lactamases by SM 7338; A Novel Carbapenem Antibacterial. 28th ICAAC, Los Angeles, October 1988. Abstract 606.
- [Background] Hamacher J, Vogel F, Lichey J, Kohl FV, Diwok K, Wendel H, Lode H. Treatment of acute bacterial exacerbations of chronic obstructive pulmonary disease in hospitalised patients--a comparison of meropenem and imipenem/cilastatin. COPD Study Group. J Antimicrob Chemother. 1995 Jul;36 Suppl A:121-33. doi: 10.1093/jac/36.suppl_a.121. PMID 8543488
- [Background] Heyland DK, Cook DJ, Griffith L, Keenan SP, Brun-Buisson C. The attributable morbidity and mortality of ventilator-associated pneumonia in the critically ill patient. The Canadian Critical Trials Group. Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 1):1249-56. doi: 10.1164/ajrccm.159.4.9807050. PMID 10194173
- [Background] Investigational Brochure, Drug Development Department, AstraZeneca Pharmaceuticals, Wilmington, Delaware 19897.
- [Background] Jones RN, Barry AL, et al. Antimicrobial Activity of SM 7338, A New DHP-1 Stable Carbapenem. 28th ICAAC, Los Angeles, October 1988. Abstract 597.
- [Background] Kayser FH, Morenzoni G. Activity of SM 7338, A New Carbapenem Antibacterial Against Gram-Positive Bacteria. 28th ICAAC, Los Angeles, October 1988. Abstract 603.
- [Background] Kollef MH, Sherman G, Ward S, Fraser VJ. Inadequate antimicrobial treatment of infections: a risk factor for hospital mortality among critically ill patients. Chest. 1999 Feb;115(2):462-74. doi: 10.1378/chest.115.2.462. PMID 10027448
- [Background] Kollef MH, Silver P, Murphy DM, Trovillion E. The effect of late-onset ventilator-associated pneumonia in determining patient mortality. Chest. 1995 Dec;108(6):1655-62. doi: 10.1378/chest.108.6.1655. PMID 7497777
- [Background] Lancero MG, Young LS. In Vitro Studies with SM 7338; A Novel Carbapenem with Broad Bactericidal Activity. 28th ICAAC, Los Angeles, October 1988. Abstract 602.
- [Background] Lode H, Hamacher J, Eller J, Schaberg T. Changing role of carbapenems in the treatment of lower respiratory tract infections. Scand J Infect Dis Suppl. 1995;96:17-23. PMID 7652498
- [Background] Luna CM, Vujacich P, Niederman MS, Vay C, Gherardi C, Matera J, Jolly EC. Impact of BAL data on the therapy and outcome of ventilator-associated pneumonia. Chest. 1997 Mar;111(3):676-85. doi: 10.1378/chest.111.3.676. PMID 9118708
- [Background] McEachern R, Campbell GD Jr. Hospital-acquired pneumonia: epidemiology, etiology, and treatment. Infect Dis Clin North Am. 1998 Sep;12(3):761-79, x. doi: 10.1016/s0891-5520(05)70209-9. PMID 9779389
- [Background] Meduri GU, Chastre J. The standardization of bronchoscopic techniques for ventilator-associated pneumonia. Chest. 1992 Nov;102(5 Suppl 1):557S-564S. doi: 10.1378/chest.102.5_supplement_1.557s. No abstract available. PMID 1424930
- [Background] Moellering RC Jr, Eliopoulos GM, Sentochnik DE. The carbapenems: new broad spectrum beta-lactam antibiotics. J Antimicrob Chemother. 1989 Sep;24 Suppl A:1-7. doi: 10.1093/jac/24.suppl_a.1. PMID 2681123
- [Background] Neu HG, Saha G, Chin NX. In Vitro Activity of SM 7338; A New Carbapenem, Compared with Other Antibacterials Against Multiply Resistant Bacteria. 28th ICAAC, Los Angeles, October 1988. Abstract 601.
- [Background] Nord CE, Lindmark A, Persson I. Susceptibility of Anaerobic Bacteria to SM 7338. 28th ICAAC, Los Angeles, October 1988. Abstract 596.
- [Background] Okuda T, Fukasawa M, Tanio T, et al. SM 7338, A New Carbapenem Antibacterial: In Vitro and In Vivo Antibacterial Activities. 27th ICAAC, New York, October 1987. Abstract 757.
- [Background] Quinn JP, Studemeister AE, DiVincenzo CA, Lerner SA. Resistance to imipenem in Pseudomonas aeruginosa: clinical experience and biochemical mechanisms. Rev Infect Dis. 1988 Jul-Aug;10(4):892-8. doi: 10.1093/clinids/10.4.892. PMID 3142013
- [Background] Sanford Guide to Antimicrobial Therapy. Thirty-third Edition, 2003. Gilbert DN, Moellering RC, Sande MA.
- [Background] Scheld WM, Mandell GL. Nosocomial pneumonia: pathogenesis and recent advances in diagnosis and therapy. Rev Infect Dis. 1991 Jul-Aug;13 Suppl 9:S743-51. doi: 10.1093/clinids/13.supplement_9.s743. PMID 1925319
- [Background] Slaney L, Chubb H, Mohammed Z, et al. In Vitro Activity of SM 7338 Against Neisseria gonorrhoeae (Gc), Haemophilus ducreyi (Hd) and Haemophilus influenzae. 28th ICAAC, Los Angeles, October 1988. Abstract 604.
- [Background] Strasbaugh LJ. Nosocomial repiratory infections. In: Mandell GL, Bennett JE, Dolin R, editors. Principles and practice of infectious disease. Philadelphia: Churchill Livingstone, 2000: 3021-3026.
- [Background] Sumita Y, Fukasawa M, Okunda T. SM 7338, A New Carbapenem Antibacterial: Affinities for PBP's and Morphological Changes. 27th ICAAC, New York, October 1987. Abstract 756.
- [Background] Sumita Y, Inoue M, Mitsuhashi S. In Vitro Antibacterial Activity of SM 7338. 28th ICAAC, Los Angeles, October 1988. Abstract 600.
- [Background] Sunagawa M, Matsumura H, Inoue T, et al. SM 7338, A New Carbapenem Antibacterial: Structure-Activity Relations and Physiochemical Properties. 27th ICAAC, New York, October 1987. Abstract 752.
- [Background] TALKE H, SCHUBERT GE. [ENZYMATIC UREA DETERMINATION IN THE BLOOD AND SERUM IN THE WARBURG OPTICAL TEST]. Klin Wochenschr. 1965 Feb 1;43:174-5. doi: 10.1007/BF01484513. No abstract available. German. PMID 14258517
- [Background] Torres A, Aznar R, Gatell JM, Jimenez P, Gonzalez J, Ferrer A, Celis R, Rodriguez-Roisin R. Incidence, risk, and prognosis factors of nosocomial pneumonia in mechanically ventilated patients. Am Rev Respir Dis. 1990 Sep;142(3):523-8. doi: 10.1164/ajrccm/142.3.523. PMID 2202245
- [Background] Torres A, Bauer TT, Leon-Gil C, Castillo F, Alvarez-Lerma F, Martinez-Pellus A, Leal-Noval SR, Nadal P, Palomar M, Blanquer J, Ros F. Treatment of severe nosocomial pneumonia: a prospective randomised comparison of intravenous ciprofloxacin with imipenem/cilastatin. Thorax. 2000 Dec;55(12):1033-9. doi: 10.1136/thorax.55.12.1033. PMID 11083889
- [Background] Trouillet JL, Chastre J, Vuagnat A, Joly-Guillou ML, Combaux D, Dombret MC, Gibert C. Ventilator-associated pneumonia caused by potentially drug-resistant bacteria. Am J Respir Crit Care Med. 1998 Feb;157(2):531-9. doi: 10.1164/ajrccm.157.2.9705064. PMID 9476869
- [Background] Vetter N. The Use of Meropenem ('Merrem'/'Meronen') in the Therapy of Hospital-acquired Lower Respiratory Infections: a Review of Clinical Experience. 18th International Congress of Chemotherapy, Stockholm, Sweden, 27 June-2 July, 1993. Abstract 70.
- [Background] Wise R, Andrews JM, Ashby JP. The Bactericidal Activity of the Carbapenem, SM 7338, Alone and in Combination. 28th ICAAC, Los Angeles, October 1988. Abstract 605.
- [Background] World Health Organization. Draft Global Strategy for the Containment of Antimicrobial Resistance. Available on the Internet at http://www.who.int/emc/amr.htm
- [Derived] Drusano GL, Corrado ML, Girardi G, Ellis-Grosse EJ, Wunderink RG, Donnelly H, Leeper KV, Brown M, Malek T, Hite RD, Ferrari M, Djureinovic D, Kollef MH, Mayfield L, Doyle A, Chastre J, Combes A, Walsh TJ, Dorizas K, Alnuaimat H, Morgan BE, Rello J, Mazo CA, Jones RN, Flamm RK, Woosley L, Ambrose PG, Bhavnani S, Rubino CM, Bulik CC, Louie A, Vicchiarelli M, Berman C. Dilution Factor of Quantitative Bacterial Cultures Obtained by Bronchoalveolar Lavage in Patients with Ventilator-Associated Bacterial Pneumonia. Antimicrob Agents Chemother. 2017 Dec 21;62(1):e01323-17. doi: 10.1128/AAC.01323-17. Print 2018 Jan. PMID 29038277

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We had 8 clinical sites: recruitment into the study began September 2010 and ended April 10, 2015.
Pre-assignment Details: Enrolled participants were excluded from the trial before assignment to groups because participants had no qualifying organisms; this includes participants with no growth on screening BAL, those with < 104 CFU/mL on BAL, and those with only Gram-positive bacteria cultured from the BAL.
Groups:
- IV Meropenem; Parenteral Aminoglycoside: Subjects assigned to this group will receive:
  * IV meropenem (2 g infused over 3 hrs q 8 hr);
  * a parenteral aminoglycoside (tobramycin or gentamicin-5mg/kg IV Q24h or amikacin 20 mg/kg IV Q24h)
  * tobramycin nebulization
  Linezolid or vancomycin (per institutional guidelines) will be available for MRSA coverage to treat potential Gram-positive pathogens.
  IV meropenem: Subjects assigned to this group will receive IV meropenem (2 g infused over 3 hrs q 8 hr).
  Parenteral aminoglycoside; tobramycin for injection USP OR gentamicin sulfate injection solution concentrate 5mg.kg IV q24h; amikacin sulfate injection USP 20 mg/kg IV q24h: a parenteral aminoglycoside (tobramycin or gentamicin-5mg/kg IV Q24h or amikacin 20 mg/kg IV Q24h)
  Linezolid or Vancomcin (per institutional guidelines) will be available for MRSA coverage.: Linezolid or vancomycin (per institutional guidelines) will be available for MRSA coverage.
  tobramycin nebulization: tobramycin nebulization 600mg/day
- I.V. Meropenem: Subjects assigned to this group will receive IV meropenem (2 g infused over 3 hrs q 8 hr).
  Linezolid or vancomycin (per institutional guidelines) will be available for MRSA coverage to treat Gram-positive pathogens.
  **NOTE: Empiric MRSA coverage is allowed in both arms. This therapy is advised for any subjects with known or suspected MRSA entering the study. Once microbiologic results are available, this coverage may be discontinued at the investigator's discretion.
  I.V. Meropenem: Subjects assigned to this group will receive IV meropenem (2 g infused over 3 hrs q 8 hr).
  Linezolid or vancomycin (per institutional guidelines) will be available for MRSA coverage
  Linezolid or Vancomcin (per institutional guidelines) will be available for MRSA coverage.: Linezolid or vancomycin (per institutional guidelines) will be available for MRSA coverage.
Period: Overall Study
Arm/Group | IV Meropenem; Parenteral Aminoglycoside | I.V. Meropenem
Started | 13 | 30
Completed | 6 | 17
Not Completed | 7 | 13
Not completed — no qualifying organism | 6 | 12
Not completed — changed to palliative care | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Number of patients enrolled in the study and who had a baseline BAL.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Meropenem; Parenteral Aminoglycoside | I.V. Meropenem | Total
Number analyzed (Participants) | 13 | 30 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 20 | 26
  >=65 years | 7 | 10 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (18.3) | 58.4 (12.6) | 59.2 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 6 | 17 | 23
Region of Enrollment [Number; unit: participants]
  United States | 11 | 18 | 29
  France | 2 | 11 | 13
  Spain | 0 | 1 | 1
Baseline acute physiology and chronic health evaluation II (APACHE II) score [Mean (Standard Deviation); unit: units on a scale] — A severity of disease classification system applied within 24 hours of patient admission to an ICU. The point score is calculated from a patient's age and physiological measurements. The range of score is between 0-71. Physiological measurements and all ages fit into that range. Note: the higher the score, the higher the probability of death.
  units on a scale | 22.6 (4.6) | 21.0 (6.2) | 21.5 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Suppression and Emergence of Resistance
Description: The emergence of resistance is defined as a change of meropenem MIC or aminoglycoside MIC by two tube dilutions (fourfold) from baseline when assessed at the second BAL procedure on day 5/early extubation. Patients are evaluable for this endpoint IF they had baseline BAL and Day 5/early extubation and if they had positive cultures on baseline and Day/EE.
Time Frame: up to 28 days after enrollment
Population: All patients in the ME population with BAL at baseline and at Day 5/EE and pathogens collected at baseline BAL and at Day 5/EE BAL.
Measure: Number; unit: participants
Arm/Group | IV Meropenem; Parenteral Aminoglycoside | I.V. Meropenem
Number analyzed (Participants) | 0 | 6
participants
  suppression of emergence of resistance |  | 5
  emergence of resistance |  | 1

2. Secondary Outcome: Clinical Response
Description: Percentage of patients with successful responses by efficacy endpoint, treatment group and population (n/N)
Time Frame: End of treatment - up to 28 days after enrollment
Population: The ME population, 19 subjects were analyzed and the m-MITT population, 24 were analyzed. Not all subjects were evaluable for each endpoint.
Measure: Count of Participants; unit: Participants
Groups:
- ME Group - Meropenem Plus Aminoglycoside; MEGroup - Meropenem Only: Percentage of patients with successful responses by efficacy endpoint, Microbiologic Evaluable (ME) group and population
- m-MITT Group - Meropenem Plus Aminoglycoside; m-MITT Group - Meropenem Only: Percentage of patients with successful responses by efficacy endpoint, Microbiologically modified ITT (m-MITT) group and population.
Arm/Group | ME Group - Meropenem Plus Aminoglycoside | MEGroup - Meropenem Only | m-MITT Group - Meropenem Plus Aminoglycoside | m-MITT Group - Meropenem Only
Number analyzed (Participants) | 4 | 15 | 6 | 18
Participants | 2 | 8 | 2 | 8

3. Secondary Outcome: Clinical Response in Subjects Who Received Prior Antibiotics
Description: Percentage of patients with successful responses by efficacy endpoint, treatment group and population (n/N)
Time Frame: End of treatment - up to 28 days after enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- ME Group - Meropenem Only: Percentage of patients with successful responses by efficacy endpoint, Microbiologic Evaluable (ME) group and population.
Arm/Group | ME Group - Meropenem Plus Aminoglycoside | ME Group - Meropenem Only | m-MITT Group - Meropenem Plus Aminoglycoside | m-MITT Group - Meropenem Only
Number analyzed (Participants) | 3 | 5 | 4 | 6
Participants | 1 | 2 | 1 | 2

4. Secondary Outcome: Overall Microbiologic Response
Description: Percentage of patients with successful responses by efficacy endpoint, treatment group and population (n/N)
Time Frame: End of treatment - up to 28 days after enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ME Group - Meropenem Plus Aminoglycoside | ME Group - Meropenem Only | m-MITT Group - Meropenem Plus Aminoglycoside | m-MITT Group - Meropenem Only
Number analyzed (Participants) | 4 | 15 | 6 | 18
Participants | 2 | 6 | 2 | 7

5. Secondary Outcome: Pretreatment Pathogen Response
Description: Percentage of patients with successful responses by efficacy endpoint, treatment group and population (n/N)
Time Frame: End of treatment - up to 28 days after enrollment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ME Group - Meropenem Plus Aminoglycoside | ME Group - Meropenem Only | m-MITT Group - Meropenem Plus Aminoglycoside | m-MITT Group - Meropenem Only
Number analyzed (Participants) | 4 | 15 | 6 | 18
Participants | 3 | 9 | 3 | 11

6. Secondary Outcome: Suppression of the Emergence of Resistance in Other Gram-negative Pathogens
Description: Percentage of patients with successful responses by efficacy endpoint, treatment group and population (n/N)
Time Frame: Day 5/Early Extubation
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ME Group - Meropenem Plus Aminoglycoside | ME Group - Meropenem Only | m-MITT Group - Meropenem Plus Aminoglycoside | m-MITT Group - Meropenem Only
Number analyzed (Participants) | 1 | 1 | 1 | 2
Participants | 1 | 1 | 1 | 2

7. Secondary Outcome: Occurrence of Repeat Negative Cultures
Description: Percentage of patients with successful responses by efficacy endpoint, treatment group and population (n/N)
Time Frame: Day 5/Early Extubation
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ME Group - Meropenem Plus Aminoglycoside | ME Group - Meropenem Only | m-MITT Group - Meropenem Plus Aminoglycoside | m-MITT Group - Meropenem Only
Number analyzed (Participants) | 4 | 15 | 4 | 17
Participants | 3 | 6 | 3 | 7

8. Secondary Outcome: Mortality
Description: Percentage of patients who died by efficacy endpoint, treatment group and population (n/N)
Time Frame: 14 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ME Group - Meropenem Plus Aminoglycoside | ME Group - Meropenem Only | m-MITT Group - Meropenem Plus Aminoglycoside | m-MITT Group - Meropenem Only
Number analyzed (Participants) | 4 | 15 | 6 | 18
Participants | 1 | 0 | 2 | 2

9. Secondary Outcome: Mortality
Description: Percentage of patients who died by efficacy endpoint, treatment group and population (n/N)
Time Frame: 28 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ME Group - Meropenem Plus Aminoglycoside | ME Group - Meropenem Only | m-MITT Group - Meropenem Plus Aminoglycoside | m-MITT Group - Meropenem Only
Number analyzed (Participants) | 4 | 15 | 6 | 18
Participants | 2 | 1 | 3 | 3

ADVERSE EVENTS:
Arm/Group | IV Meropenem; Parenteral Aminoglycoside | I.V. Meropenem
Serious Adverse Events (participants affected / at risk) | 6/13 | 11/30
Other Adverse Events (participants affected / at risk) | 0/13 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Meropenem; Parenteral Aminoglycoside (N=13) | I.V. Meropenem (N=30)
cutaneous eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
reinforced duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
pneomonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
COPD with acute exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Note: this patient in group 2 (IV mero only) experienced 2 SAES that occurred in separate organ systems: AICD fired/NSTEMI and COPD with acute exacerbation. Therefore, this patient was counted twice.
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
AICD fired/NSTEMI (Cardiac disorders) | 0 (0) | 1 (1) — Note: this patient in group 2 (IV mero only) experienced 2 SAES that occurred in separate organ systems: AICD fired/NSTEMI and COPD with acute exacerbation. Therefore, this patient was counted twice.
PEA arrest (Cardiac disorders) | 1 (1) | 0 (0)
multi-organ failure (General disorders) | 0 (0) | 2 (2)
multi-organ failure due to distributive and cardiogenic shock (General disorders) | 1 (1) | 0 (0)
stroke (General disorders) | 0 (0) | 1 (1) — Note: this patient in group 2 (IV mero only) experienced 2 SAES that occurred in separate organ systems: Pulmonary embolism and stroke.. Therefore, this patient was counted twice.
pulmonary embolism (General disorders) | 0 (0) | 1 (1) — Note: this patient in group 2 (IV mero only) experienced 2 SAES that occurred in separate organ systems: Pulmonary embolism and stroke. Therefore, this patient was counted twice.
refractory shock (General disorders) | 0 (0) | 1 (1)
septic shock (General disorders) | 0 (0) | 1 (1)
cardiorespiratory arrest (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days